CLINICAL TRIAL: NCT07166432
Title: Development, Application, and Mechanistic Investigation of a Novel Minimally-Invasive Bidirectional Epidural Cerebellar Stimulation Technique for Cerebellar Cognitive Affective Syndrome
Status: Recruiting | Type: Observational
Sponsor: Peking University First Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: PKUFH-URO-CCAS-2025-MI-BES
Record Dates: First submitted 2025-09-03; First posted 2025-09-10 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-06

CONDITIONS: Cerebellar Atrophy; Etiology; Physiopathology

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: observational diagnostic model development — observational diagnostic model development

SUMMARY:
Building on previous findings regarding microglial immune function and the immunosuppressive effects of glucocorticoids, this project centers on the cerebellum's role in cognitive science. Using Cushing's syndrome-induced cerebellar atrophy leading to CCAS as a model, we aim to elucidate the pathogenic mechanisms governed by the neuro-adrenal-immune network and to uncover the molecular basis by which a novel minimally invasive brain-machine fusion system ameliorates cerebellar ataxia and cognitive impairment.

ELIGIBILITY:
Inclusion Criteria:

* 1. Clinically and biochemically confirmed ACTH-dependent or ACTH-independent Cushing syndrome (loss of serum cortisol circadian rhythm, elevated 24-hour urinary free cortisol, and failure to suppress on low-dose dexamethasone suppression test).

  2. Cranial MRI demonstrating unequivocal cerebellar atrophy (CCAS imaging criterion: cerebellar hemisphere or vermian volume ≥1.5 SD below age-matched normative data).

  3. Established clinical diagnosis of CCAS (meets Schmahmann criteria, CCAS-S total score ≥20).

  4. Cerebellar ataxia rating scale (SARATA) ≥10, indicating at least moderate motor ataxia.

  5. Positive cognitive impairment screen (MoCA <26, or Z-scores ≤-1.5 in at least two cognitive domains).

  6. Willingness to undergo minimally invasive epidural cerebellar stimulation and provision of written informed consent.

Exclusion Criteria:

Patients with significant systemic disease; occurrence of major complications or irreproducible, critical deviations in data collection or experimental procedures; or any circumstance rendering continued participation inappropriate-including clinical deterioration, serious adverse events, or poor compliance-will result in discontinuation of the subject's enrollment.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged 18-80 years who have documented hypercortisolism (Cushing syndrome) on clinical testing and are assessed as having decision-making capacity.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-06-28 (Actual); Primary Completion 2028-06-01 (Estimated); Study Completion 2028-06-01 (Estimated)

PRIMARY OUTCOMES:
A "dual clinical response" at 12 weeks post-treatment, defined as a ≥5-point improvement in the Cerebellar Cognitive Affective Syndrome Scale (CCAS-S) total score AND a ≥6-point improvement in the Scale for Assessment and Rating of Ataxia (SARATA) total | from 2025 to 2028

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Urology, Peking University First Hospital, Beijing, 100034, Beijing, China